CLINICAL TRIAL: NCT03391661
Title: Openness to Cognitive Approach of Nonspecific Chronic Pain
Brief Title: University of Michigan / Wayne State Chronic Pain Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Distinguished Professor of Psychology, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00121358
Record Dates: First submitted 2017-12-22; First posted 2018-01-05 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Chronic Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Pain and the Brain (Experimental): This condition is a 15 to 20-minute exercise that patients complete in which they examine variables in themselves that suggest that their pain is driven by central nervous system processes / their brains.
  Interventions: Behavioral: Pain neuroscience education patient exercise
- Health Behavior Control (Placebo Comparator): This 15 to 20-minute exercise is designed as a control condition that has face validity as helpful and that relates to health. Thus, patients are asked to examine various domains of their own health behavior as engaged in over the past 24 hours (e.g., nutrition, sleep, exercise, hygiene, social connections).
  Interventions: Behavioral: Health behavior control intervention

INTERVENTIONS:
Behavioral: Pain neuroscience education patient exercise — Patients complete a 15 to 20-minute on-line exercise that inquires about 5 domains: the degree of central sensitization symptoms, catastrophizing and kinesiophobia, personality factors, stressors that triggered or exacerbated the pain, and adverse childhood experiences.
  Arms: Chronic Pain and the Brain
Behavioral: Health behavior control intervention — Patients engage in a 15 to 20-minute on-line exercise examining their health behaviors in five domains: exercise, sleep, diet, hygiene, and social connections.
  Arms: Health Behavior Control

SUMMARY:
This study is designed to determine if a brief educational program can alter the attitudes and knowledge of individuals with chronic back pain, which is likely to be non-structural in nature.

Individuals will be randomly assigned to an experimental condition (performs written educational and emotional awareness exercises) or a control condition (completes a general health activities questionnaire). Comparisons will be made to assess the degree of centralized pain features and functional improvements at 1-month follow-up. A 10-month follow-up as a secondary endpoint is also planned.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults ages 18 years or older with internet access who are referred to the University of Michigan Health Service Physical Medicine and Rehabilitation Spine Program identified the physician with chronic nonspecific back pain (longer than 3 months) or fibromyalgia. Degenerative changes seen on imaging are considered nonspecific. Alternatively, enrolled in the University of Michigan Health Research Volunteer Pool with a profile that includes chronic low back pain or fibromyalgia.

Exclusion Criteria:

* Any signs of a serious underlying condition (cancer, infection, cauda equine), spinal stenosis or radiculopathy, or other specific spinal cause (vertebral compression fracture or ankylosing spondylitis). Those patients who are being considered for an interventional spine procedures or surgical consults would not be included in this study.
* Individuals receiving or applying for compensation or disability, the inability to provide written informed consent, severe physical impairment (e.g. blindness, deafness), co-morbid medical condition limiting function (e.g. malignant cancer), the use of illicit drug use, or a psychiatric condition that would limit judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | Change from baseline to 1-Month follow-up (with secondary 10-month follow-up)
  Self-reported pain and dysfunction

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System: Depression short form 8b | Change from baseline to 1-Month follow-up (with secondary 10-month follow-up)
  Self-reported depression
Patient-Reported Outcomes Measurement Information System: Anxiety short form 8a | Change from baseline to 1-Month follow-up (with secondary 10-month follow-up)
  Self-reported anxiety
Patient-Reported Outcomes Measurement Information System: Anger short form 5a | Change from baseline to 1-Month follow-up (with secondary 10-month follow-up)
  Self-reported anger
Pain attributions questionnaires | Change from baseline to 1-Month follow-up (with secondary 10-month follow-up)
  Two self-report questionnaires were developed to assess psychological and brain influences on pain. The 4-item psychological attribution scale assesses patients' beliefs that their thoughts and feelings and psychological therapy impacts pain, and the 3-item brain attribution scale assesses patient's beliefs that their pain is brain-based. Mean scores will be computed for both scales separately (0-4; higher scores indicating greater belief that pain is a brain-related [brain attribution] construct and that pain is affected by thoughts, feelings, and psychological interventions [psychological attribution])
Pain Stages of Change Questionnaire | Change from baseline to 1-Month follow-up (with secondary 10-month follow-up)
  The Pain Stages of Change questionnaire (Kerns, Rosenberg, Jamison, Caudill, & Haythornthwaite, 1997): an overall readiness score will be calculated using mean scores of the four subscales. Readiness is the sum of patient mean ratings for contemplation (C; 1-5), action (A; 1-5), and maintenance (M; 1-5), minus the mean score for precontemplation (PC; 1-5): C + A + M - PC = Readiness. Higher scores indicate greater readiness.
Pain Catastrophizing Scale | Change from baseline to 1-Month follow-up (with secondary 10-month follow-up)
  Pain Catastrophizing Scale (Sullivan et al., 1995): A summed score of the 13 catastrophizing items will be computed (0-52, higher scores indicate greater catastrophizing)
Tampa Scale for Kinesiophobia | Change from baseline to 1-Month follow-up (with secondary 10-month follow-up)
  The Tampa Kinesiophobia Scale (Miller, Kori, &Todd, 1991): A mean score of the 11 items will be computed (1-4, higher scores indicating greater kinesiophobia)
Satisfaction with Life Scale | Change from baseline to 1-month follow-up (with secondary 10-month follow-up)
  The Satisfaction with Life Scale (Emmons, Larsen, & Griffin, 1985): A mean score of the 5 items will be computed (1-7, higher scores indicating greater life satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: David Kohns, MD, Principal Investigator — University of Michigan; Mark A Lumley, PhD, Study Director — Wayne State University
Locations (1):
- University of Michigan Physical Medicine and Rehabilitation Department, Ann Arbor, Michigan, United States